CLINICAL TRIAL: NCT04552678
Title: Healthy Bodies Project: Modifying Family and Preschool Environments to Prevent Obesity
Brief Title: Healthy Bodies Project to Prevent Childhood Obesity
Acronym: Healthy Bodies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Lori Francis, Associate Professor of Biobehavioral Health, Penn State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-68001-23233
Record Dates: First submitted 2020-09-07; First posted 2020-09-17 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Obesity, Childhood
Keywords: nutrition knowledge; food literacy; physical activity; executive function; emotion regulation; eating regulation; parenting; food parenting
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Emotional Regulation | interventions — Diet, Healthy

STUDY DESIGN:
Intervention Model Description: The study utilizes a 2x4 factorial design with 16 conditions. Classrooms are the unit of randomization. Classrooms are randomized into 1 of 16 conditions that vary based on whether or not the following treatments are turned on or off: Healthy Eating Classroom Curriculum; Active Play Classroom Curriculum; Self-Regulation Classroom Curriculum; Enhanced Parent Education. All classrooms receive a Food Literacy curriculum.
Who Masked: Outcomes Assessor
Masking Description: Assessors who collect data from children are blind to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Healthy Eating, Active Play, Self-Regulation, Parent Education (Experimental): Classrooms receive all curricula (Food Literacy, Healthy Eating, Active Play, Self-Regulation Curriculum) and Parent Education
  Interventions: Behavioral: Healthy Eating, Active Play, Self-Regulation, Parent Education
- Healthy Eating, Active Play, Self-Regulation (Experimental): Classrooms receive all curricula (Food Literacy, Healthy Eating, Active Play, Self-Regulation Curriculum), but no Parent Education
  Interventions: Behavioral: Healthy Eating, Active Play, Self-Regulation
- Healthy Eating, Active Play, Parent Education (Experimental): Classrooms receive the core Food Literacy Curriculum, the Healthy Eating Curriculum, the Active Play Curriculum, and Parent Education
  Interventions: Behavioral: Healthy Eating, Active Play, Parent Education
- Healthy Eating + Active Play (Experimental): Classrooms receive the core Food Literacy Curriculum, the Healthy Eating Curriculum, the Active Play Curriculum, but no Parent Education
  Interventions: Behavioral: Healthy Eating + Active Play
- Healthy Eating, Self-Regulation, Parent Education (Experimental): Classrooms receive the core Food Literacy Curriculum, the Healthy Eating Curriculum, the Self-Regulation Curriculum, and Parent Education
  Interventions: Behavioral: Healthy Eating, Self-Regulation, Parent Education
- Healthy Eating + Self-Regulation (Experimental): Classrooms receive the core Food Literacy Curriculum, the Healthy Eating Curriculum, the Self-Regulation Curriculum, but no Parent Education
  Interventions: Behavioral: Healthy Eating + Self-Regulation
- Healthy Eating + Parent Education (Experimental): Classrooms receive the core Food Literacy Curriculum, the Healthy Eating Curriculum, and Parent Education
  Interventions: Behavioral: Healthy Eating + Parent Education
- Healthy Eating Only (Experimental): Classrooms receive the core Food Literacy Curriculum, the Healthy Eating Curriculum, but no Parent Education
  Interventions: Behavioral: Healthy Eating Only
- Active Play, Self-Regulation, Parent Education (Experimental): Classrooms receive the core Food Literacy Curriculum, the Active Play Curriculum, the Self-Regulation Curriculum, and Parent Education
  Interventions: Behavioral: Active Play, Self-Regulation, Parent Education
- Active Play + Self-Regulation (Experimental): Classrooms receive the core Food Literacy Curriculum, the Active Play Curriculum, the Self-Regulation Curriculum, but no Parent Education
  Interventions: Behavioral: Active Play + Self-Regulation
- Active Play + Parent Education (Experimental): Classrooms receive the core Food Literacy Curriculum, the Active Play Curriculum, and Parent Education
  Interventions: Behavioral: Active Play + Parent Education
- Active Play Only (Experimental): Classrooms receive the core Food Literacy Curriculum, the Active Play Curriculum, but no Parent Education
  Interventions: Behavioral: Active Play Only
- Self-Regulation + Parent Education (Experimental): Classrooms receive the core Food Literacy Curriculum, the Self-Regulation Curriculum, and Parent Education
  Interventions: Behavioral: Self-Regulation + Parent Education
- Self-Regulation Only (Experimental): Classrooms receive the core Food Literacy Curriculum, the Self-Regulation Curriculum, but no Parent Education
  Interventions: Behavioral: Self-Regulation Only
- Food Literacy + Parent Education (Experimental): Classrooms receive the core Food Literacy Curriculum, and parents are invited to complete web-based education modules.
  Interventions: Behavioral: Food Literacy + Parent Education
- Food Literacy Only (Experimental): Classrooms only receive the core Food Literacy Curriculum, and no other intervention materials or parent education.
  Interventions: Behavioral: Food Literacy Only

INTERVENTIONS:
Behavioral: Healthy Eating, Active Play, Self-Regulation, Parent Education — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Healthy Eating curriculum, an 11-lesson Active Play curriculum, and an 11-lesson Self-Regulation curriculum. Parents will receive access to web-based resources on food literacy, and will be invited to complete 18 web-based education modules on topics including improving household routines, managing children's behaviors and emotions, improving children's sleep patterns, improving access to healthy foods, healthy meal and snack preparation, modeling healthy eating and activity behaviors, and improving family activity patterns.
  Arms: Healthy Eating, Active Play, Self-Regulation, Parent Education
Behavioral: Healthy Eating, Active Play, Self-Regulation — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Healthy Eating curriculum, an 11-lesson Active Play curriculum, and an 11-lesson Self-Regulation curriculum. Parents will receive access to web-based resources on food literacy.
  Arms: Healthy Eating, Active Play, Self-Regulation
Behavioral: Healthy Eating, Active Play, Parent Education — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Healthy Eating curriculum, and an 11-lesson Active Play curriculum. Parents will receive access to web-based resources on food literacy, and will be invited to complete 18 web-based education modules on topics including improving household routines, managing children's behaviors and emotions, improving children's sleep patterns, improving access to healthy foods, healthy meal and snack preparation, modeling healthy eating and activity behaviors, and improving family activity patterns.
  Arms: Healthy Eating, Active Play, Parent Education
Behavioral: Healthy Eating + Active Play — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Healthy Eating curriculum, and an 11-lesson Active Play curriculum. Parents will receive access to web-based resources on food literacy.
  Arms: Healthy Eating + Active Play
Behavioral: Healthy Eating, Self-Regulation, Parent Education — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Healthy Eating curriculum, and an 11-lesson Self-Regulation curriculum. Parents will receive access to web-based resources on food literacy, and will be invited to complete 18 web-based education modules on topics including improving household routines, managing children's behaviors and emotions, improving children's sleep patterns, improving access to healthy foods, healthy meal and snack preparation, modeling healthy eating and activity behaviors, and improving family activity patterns.
  Arms: Healthy Eating, Self-Regulation, Parent Education
Behavioral: Healthy Eating + Self-Regulation — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Healthy Eating curriculum, and an 11-lesson Self-Regulation curriculum. Parents will receive access to web-based resources on food literacy.
  Arms: Healthy Eating + Self-Regulation
Behavioral: Healthy Eating + Parent Education — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Healthy Eating curriculum. Parents will receive access to web-based resources on food literacy, and will be invited to complete 18 web-based education modules on topics including improving household routines, managing children's behaviors and emotions, improving children's sleep patterns, improving access to healthy foods, healthy meal and snack preparation, modeling healthy eating and activity behaviors, and improving family activity patterns.
  Arms: Healthy Eating + Parent Education
Behavioral: Healthy Eating Only — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Healthy Eating curriculum. Parents will receive access to web-based resources on food literacy.
  Arms: Healthy Eating Only
Behavioral: Active Play, Self-Regulation, Parent Education — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Active Play curriculum, and an 11-lesson Self-Regulation curriculum. Parents will receive access to web-based resources on food literacy, and will be invited to complete 18 web-based education modules on topics including improving household routines, managing children's behaviors and emotions, improving children's sleep patterns, improving access to healthy foods, healthy meal and snack preparation, modeling healthy eating and activity behaviors, and improving family activity patterns.
  Arms: Active Play, Self-Regulation, Parent Education
Behavioral: Active Play + Self-Regulation — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Active Play curriculum, and an 11-lesson Self-Regulation curriculum. Parents will receive access to web-based resources on food literacy.
  Arms: Active Play + Self-Regulation
Behavioral: Active Play + Parent Education — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Active Play curriculum. Parents will receive access to web-based resources on food literacy, and will be invited to complete 18 web-based education modules on topics including improving household routines, managing children's behaviors and emotions, improving children's sleep patterns, improving access to healthy foods, healthy meal and snack preparation, modeling healthy eating and activity behaviors, and improving family activity patterns.
  Arms: Active Play + Parent Education
Behavioral: Active Play Only — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Active Play curriculum. Parents will receive access to web-based resources on food literacy.
  Arms: Active Play Only
Behavioral: Self-Regulation + Parent Education — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Self-Regulation curriculum. Parents will receive access to web-based resources on food literacy, and will be invited to complete 18 web-based education modules on topics including improving household routines, managing children's behaviors and emotions, improving children's sleep patterns, improving access to healthy foods, healthy meal and snack preparation, modeling healthy eating and activity behaviors, and improving family activity patterns.
  Arms: Self-Regulation + Parent Education
Behavioral: Self-Regulation Only — In addition to a 27-lesson, core food literacy curriculum that children across all conditions will receive, children in this condition will also be exposed to an 11-lesson Self-Regulation curriculum. Parents will receive access to web-based resources on food literacy.
  Arms: Self-Regulation Only
Behavioral: Food Literacy + Parent Education — Children in this condition will only receive a 27-lesson, core food literacy curriculum (children across all conditions will receive this curriculum). Parents will receive access to web-based resources on food literacy, and will be invited to complete 18 web-based education modules on topics including improving household routines, managing children's behaviors and emotions, improving children's sleep patterns, improving access to healthy foods, healthy meal and snack preparation, modeling healthy eating and activity behaviors, and improving family activity patterns.
  Arms: Food Literacy + Parent Education
Behavioral: Food Literacy Only — Children in this condition will only receive a 27-lesson, core food literacy curriculum (children across all conditions will receive this curriculum). Parents will receive access to web-based resources on food literacy.
  Arms: Food Literacy Only

SUMMARY:
The goal of this study is to evaluate components of a preschool-based intervention designed to (1) increase children's nutrition knowledge, (2) increase physical activity in childcare settings, (3) increase emotional, behavioral and eating-related regulation, and (4) provide guidance to parents/caregivers about appropriate parenting and child-feeding strategies that promote healthy eating behaviors, dietary patterns and physical activity in preschool-aged children. The long-term goal is to help children develop healthy habits that reduce risk for obesity.

DETAILED DESCRIPTION:
Findings from intervention studies designed to prevent obesity among preschool children are mixed. One approach to stemming the development of obesity in childhood is to alter children's choices and environments in ways that promote food literacy, acceptance of healthy foods, physical activity and self-regulation. Research on factors that influence the development of obesity in children has identified factors in children's environments that are potential targets for prevention programs. The goal of this study is to evaluate the efficacy of components designed for a preschool-based approach to preventing obesity in children. Using an innovative approach to optimizing behavioral interventions, the multiphase optimization strategy (MOST), we will examine the effects of a 28-week, randomized set of experiments designed to (1) increase children's nutrition knowledge, (2) increase physical activity in childcare settings, (3) increase emotional, behavioral and eating-related regulation, and (4) provide guidance to parents/caregivers about appropriate parenting and child-feeding strategies that promote healthy eating behaviors, dietary patterns and physical activity in preschool-aged children. Participants will include over 1300 predominantly low-income preschool children ages 3 to 5 years attending center-based childcare settings in Pennsylvania (~100 classrooms). The proposed study will provide information on the most efficacious components that produce measurable changes in children's nutrition knowledge and obesity-related behaviors. The results of this study will be used to inform the design of a randomized controlled trial to prevent obesity in children.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3 to 5 years enrolled in full-day, center-based childcare programs
* Caregiver ≥ 18 years of age
* Caregiver responsible for providing meals for child at least half of the time
* Fluent in English (caregiver and child)

Exclusion Criteria:

* Developmental delays or disorders that affect learning, mobility and eating

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2480 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Child Body Mass Index (BMI) | Change from baseline to post-assessment (5-6months) and follow-up (~9 months)
  Absolute BMI, BMI z-score (BMIz), BMI percentile (BMIp) calculated from measured height and weight
Nutrition Knowledge | Change from baseline to post-assessment (5-6months) and follow-up (~9 months)
  Ability to identify energy- vs. nutrient-dense foods using the Food Knowledge Procedure
Food Choices | Change from baseline to post-assessment (5-6months) and follow-up (~9 months)
  Children's choices between energy- vs. nutrient-dense foods for a hypothetical lunch using the Snack Selection Procedure
Physical and Sedentary Activity | Change from Baseline to Mid-Intervention (~3 months), Post-Intervention (5-6 months) and follow-up (~9 months)
  Children's engagement in sedentary and moderate-vigorous physical activity during the school day objectively measured via accelerometry.
Children's Behavioral Regulation - Observed | Change from baseline to post-assessment (5-6months) and follow-up (~9 months)
  Behavioral tasks that measure child inhibitory control: Walk a Line Slowly, Peg/Pencil Tapping Procedure and Choosing Dinky Toys.
  Assessor reports of children's emotions, attention, and behavior: Preschool Self-Regulation Assessor Report
Children's Behavioral Regulation - Parent- and Teacher-Report | Change from baseline to post-assessment (5-6months)
  Teacher reports of children's attentional focusing, impulsivity and inhibitory control: Child Behavior Questionnaire
  Parent reports of children's impulsivity and inhibitory control: Child Behavior Questionnaire
Children's Emotion Regulation - Parent- and Teacher-Report | Change from baseline to post-assessment (5-6months)
  Parent and Teacher reports of children's anger/frustration: Child Behavior Questionnaire
Children's Eating in the Absence of Hunger | Change from baseline to post-assessment (5-6months)
  Parent reported measure of children's eating in the absence of hunger due to negative emotions, fatigue/boredom, or external food cues.

SECONDARY OUTCOMES:
Children's Appetitive Behaviors | Baseline, Post-Intervention (5-6 months)
  Parent report of children's appetitive trait-like behaviors (responsiveness to food, enjoyment of food, satiety responsiveness, slowness in eating, fussiness, emotional overeating, emotional undereating, and desire for drinks). Measured using the Children's Eating Behavior Questionnaire.
Children's Food Requests | Baseline, Post-Intervention (5-6 months)
  Parental reports of children's requests for fruits, vegetables, whole grains and dairy.
Parental reports of children's requests for fruits, vegetables, whole grains and dairy | Baseline, Post-Intervention (5-6 months)
  Parent reported measure of children's eating in the absence of hunger due to negative emotions, fatigue/boredom, or external food cues.

OTHER OUTCOMES:
Food Parenting Practices | Change from baseline to post-assessment (5-6months)
  Comprehensive Feeding Practices Questionnaire to assess parental monitoring, restriction, pressure to eat, modeling, teaching about nutrition, child involvement, using food for emotional regulation, using food as a reward, child control in eating, healthy food availability, and encouraging balance. Child Feeding Questionnaire to assess child picky eating, and parents' perception of time for healthy eating.
Sociodemographics | Change from baseline to post-assessment (5-6months)
  Parent Demographic Questionnaire to assess parent age, BMI, race, education, employment, marital status and household income.
Parent Physical Activity | Change from baseline to post-assessment (5-6months)
  International Physical Activity Questionnaire (IPAQ, short form) to classify parents as sedentary, moderately active or vigorously active.
Family Media Use Patterns | Change from baseline to post-assessment (5-6months)
  Family Media Patterns questionnaire developed by the research group to measure screen use and eating during televisions viewing in children and parents.
Activity Parenting Practices | Change from baseline to post-assessment (5-6months)
  Questionnaire to measure parents' use of TV viewing as a form of family recreation, frequency of TV viewing during mealtime and children's time spent watching television (TV) or playing on computer/phone/tablet.
Child Sleep Patterns | Change from baseline to post-assessment (5-6months)
  Parent report of children's sleep duration, sleep timing and napping patterns
Food Availability, Modeling and Encouragement | Change from baseline to post-assessment (5-6months)
  Fruit and Vegetable, whole grain and dairy questionnaires, developed by the research team, to assess fruit, vegetable, whole grain and dairy availability in the home, parental encouragement to consume, and parental modeling of consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Francis, Ph.D., Principal Investigator — The Pennsylvania State University

IPD SHARING:
Plan to Share IPD: No
There is no finalized plan for which and how individual participant data will be shared. This plan will be developed in collaboration with the sponsoring institution and funders.

REFERENCES:
- See also: A child health and wellness research study funded by the U.S. Department of Agriculture (USDA) — https://sites.psu.edu/healthybodies/